CLINICAL TRIAL: NCT04318405
Title: Iron Isomaltoside 1000 in Patients With Iron Deficiency or Iron Deficiency Anemia: a Multicentric, Prospective, Longitudinal, Observational Study in Switzerland.
Brief Title: Real Life Study on Iron Isomaltoside 1000 in the Treatment of ID in CKD, Heart Failure, ObGyn, IBD, Cancer and Elective Surgery (Real-CHOICE).
Acronym: Real-CHOICE
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-PFM-2019-2654
Record Dates: First submitted 2020-03-12; First posted 2020-03-24 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Iron-Deficiency Anemia; Iron-Deficiency
Keywords: Iron isomaltoside 1000; Iron Derisomaltose 1000
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — iron isomaltoside 1000

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Iron isomaltoside 1000 — Observation of real-life treatment with iron isomaltoside 1000 / Iron Derisomaltose 1000
  Other Names: Iron Derisomaltose 1000

SUMMARY:
Real-CHOICE - designed as a prospective, longitudinal, observational, non-interventional study - will investigate the attitude of patients and physicians towards IV (intravenous) iron therapy in general and IIM (iron isomaltoside 1000) treatment particularly before and after IIM treatment in iron deficient patients with or without anemia in the real-world clinical setting after commercial availability of this product in Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* Legally capable male and female patients, aged ≥ 18 years (no upper limit);
* Written informed consent of the patient with regard to the pseudonymized documentation;
* The patients are not selected by specific inclusion or exclusion criteria, but by the indication listed in the Swiss SmPC (Summary of Product Characteristics) of Monofer®;
* Decision is taken to treat the patient with IIM in accordance with the current Swiss SmPC of Monofer® and by prescription; this decision is taken prior to and independent from the inclusion into the study.

Exclusion Criteria:

* Any contraindication regarding IIM treatment as specified in the Swiss SmPC of Monofer®;
* Retrospective observation of IIM infusion;
* Current or upcoming participation in an interventional clinical trial;
* Prior IV iron treatment or transfusion within 3 months prior to enrolment;
* Instable and/or untreated comorbidities potentially hampering the observation of the primary outcome parameter of this study;
* Prisoners or persons who are compulsorily detained (involuntarily incarcerated).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with iron deficiency (IDNA) or iron deficiency anemia (IDA) treated at the treating physician's discretion with IIM according to the Swiss SmPC for Monofer® in current practice.
Sampling Method: Non-Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Attitude of patients towards IV iron treatment evaluated with questionnaire. | Change from baseline taking into account baseline (BL) and follow-up (FU) answers. Follow-up at the latest 12 weeks after observed dosing and before a potential subsequent dosing (if available based on clinical routine follow-up).
  Rate of patients with stability or positive change in attitude.
  Questionnaire comprises the following questions:
  1. I am hesitant to be treated with IV iron.
  2. I would consider IV iron treatment due to the physician ́s choice.
  3. I would consider IV iron treatment due to its safety compared to other iron treatment options.
  4. I would consider IV iron treatment due to its efficacy compared to other iron treatment options.

SECONDARY OUTCOMES:
Effectiveness of treatment with IIM. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Iron deficiency anemia (IDA): Hb (Hemoglobin) increase ≥ 1 g/dL.
Effectiveness of treatment with IIM. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Iron deficiency without anemia (IDNA): Maintenance of baseline Hb-level and/or Hb above lower limit of normal (LLN).
Attitude of patients towards IIM treatment evaluated with questionnaire. | Complete observation time-frame (the total observation period of this study will amount to 90 months).
  Taking into account baseline (BL) and follow-up (FU) answers.
  Questionnaire comprises the following questions:
  1. I am hesitant to be treated with IIM.
  2. I would consider IIM treatment due to the physician ́s choice.
  3. I would consider IIM treatment due to its safety compared to other iron treatment options.
  4. I would consider IIM treatment due to its efficacy compared to other iron treatment options.
  5. I would consider IIM treatment due to its specific dosing and administration schedule.
Attitude of physicians towards IIM and IV iron treatment evaluated with questionnaire. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Questionnaire comprises the following questions:
  1. I am hesitant to treat with IV iron.
  2. I would consider IV iron treatment due to the patient ́s desire.
  3. I would consider IV iron treatment due to its safety compared to other iron treatment options.
  4. I would consider IV iron treatment due to its efficacy compared to other iron treatment options.
  And:
  1. I am hesitant to treat with IIM.
  2. I would consider IIM treatment due to the patient ́s desire.
  3. I would consider IIM treatment due to its safety compared to other iron treatment options.
  4. I would consider IIM treatment due to its efficacy compared to other iron treatment options.
  5. I would consider IIM treatment due to its specific dosing and administration schedule.
Patient and disease profiles at baseline. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Evaluation of kind of iron deficiency.
Patient and disease profiles at baseline. | Baseline.
  Institution of diagnosis of IDA/IDNA.
Patient and disease profiles at baseline. | Baseline.
  Etiology of iron deficiency.
Patient and disease profiles at baseline. | Baseline.
  Method of iron need determination.
Calculation of iron need based on IIM simplified dosing scheme. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Evaluation of dosing intensity of IIM.
Calculation of iron need based on IIM simplified dosing scheme. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Calculated iron need.
Calculation of iron need based on IIM simplified dosing scheme. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Determined iron need.
Calculation of iron need based on IIM simplified dosing scheme. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Difference between administered IIM dose and calculated iron need.
Treatment sequence before IIM. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Dose intensities of administration.
Treatment sequence before IIM. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Dose intervals of administration.
Reason(s) for selection of IIM. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Reasons for treatment choice of IIM in current patient populations. Reasons could be: efficacy, safety profile, quality of life, patient's preference, physician's preference, comorbidities, convenient dosing, other.
Treatment with IIM. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Dose intensity of administration.
Treatment with IIM. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Mode of administration.
Treatment with IIM. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Duration of infusion.
Treatment satisfaction of physician and patient upon treatment. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Rate of physicians and patients with stability or positive change in satisfaction upon IIM treatment.
Effectiveness of treatment with IIM: whole blood count changes. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Red blood cell count
Effectiveness of treatment with IIM: whole blood count changes. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  White blood cell count
Effectiveness of treatment with IIM: whole blood count changes. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Hemoglobin
Effectiveness of treatment with IIM: whole blood count changes. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Hematocrit
Effectiveness of treatment with IIM: whole blood count changes. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Platelets
Effectiveness of treatment with IIM: total Hb increase. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Hemoglobin
Effectiveness of treatment with IIM: serum ferritin increase. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Serum ferritin
Effectiveness of treatment with IIM: serum ferritin increase. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Transferrin saturation (TfS)
Effectiveness of treatment with IIM: serum ferritin increase. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Soluble transferrin receptor (sTfR)
Effectiveness of treatment with IIM: serum ferritin increase. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Phosphate level
Effectiveness of treatment with IIM: CRP (C-reactive protein) status. | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  CRP status.
Safety and tolerability of treatment with IIM, including frequency and severity of treatment-emergent AEs (Adverse Events) / ADRs (Adverse Drug Reactions). | Complete observation time-frame (the total observation period of this study per patient will amount to 3 months).
  Number of patients with:
  * Treatment-emergent adverse events (maximum grade per patient),
  * Grade 3/4 treatment-emergent adverse drug reactions,
  * Grade 3/4 treatment-emergent serious adverse events,
  * Treatment-emergent serious adverse drug reactions,
  * Pre-treatment adverse events,
  * Pre-treatment serious adverse events,
  * Follow-up adverse events,
  * Follow-up serious adverse events.

CONTACTS AND LOCATIONS:
Locations (21):
- Switzerland (21):
  - 21, Basel
  - 9, Basel
  - 1, Bern
  - 15, Biel
  - 19, Brugg
  - 18, Gossau
  - 11, Kreuzlingen
  - 12, Kreuzlingen
  - 8, Kreuzlingen
  - 5, Liestal
  - 20, Opfikon
  - 16, Rheinfelden
  - 13, Sankt Gallen
  - 17, Sankt Gallen
  - 7, Sion
  - 6, Spreitenbach
  - 14, Steinach
  - 10, Wettingen
  - 3, Wohlen
  - 2, Zurich
  - 4, Zurich

IPD SHARING:
Plan to Share IPD: No